CLINICAL TRIAL: NCT00391625
Title: An Open-Label Extension of Study TKT025 Evaluating Long Term Safety in Patients With Type 1 Gaucher Disease Receiving DRX008A Enzyme Replacement Therapy
Brief Title: Open-Label Extension Study Evaluating Long Term Safety in Patients With Type 1 Gaucher Disease Receiving DRX008A (ERT)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TKT025EXT
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-05

CONDITIONS: Gaucher Disease
Keywords: Gaucher disease, Enzyme Replacement Therapy
MeSH Terms: conditions — Gaucher Disease | interventions — Glucosylceramidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GA-GCB (Experimental): 15-60 U/kg every other week via intravenous infusion
  Interventions: Drug: GA-GCB

INTERVENTIONS:
Drug: GA-GCB — 15-60 U/kg every other week via intravenous infusion
  Other Names: VPRIV®; velaglucerase alfa; gene-activated glucocerebrosidase; DRX008

SUMMARY:
Gaucher disease is a rare lysosomal storage disorder caused by the deficiency of the enzyme glucocerebrosidase (GCB). Due to the deficiency of functional GCB, glucocerebroside accumulates within macrophages leading to cellular engorgement, organomegaly, and organ system dysfunction. The purpose of this study is to evaluate the long term safety of enzyme replacement therapy with DRX008A (VPRIV®, GA-GCB; velaglucerase alfa) in patients with type 1 Gaucher disease.

DETAILED DESCRIPTION:
Type 1 Gaucher disease, the most common form, accounts for more than 90% of all cases and does not involve the central nervous system (CNS). Typical manifestations of type 1 Gaucher disease include hepatomegaly, splenomegaly, thrombocytopenia, bleeding tendencies, anemia, hypermetabolism, skeletal pathology, growth retardation, pulmonary disease, and decreased quality of life. Gene-Activated® human glucocerebrosidase (the long term safety of enzyme replacement therapy with DRX008A (GA-GCB; velaglucerase alfa) is produced in a continuous human cell line using proprietary gene-activation technology and has an identical amino acid sequence to the naturally occurring human enzyme. GA-GCB (velaglucerase alfa) contains terminal mannose residues that target the enzyme to the macrophages-the primary target cells in Gaucher disease. This study was designed to evaluate the long term safety of GA-GCB (velaglucerase alfa) in patients with Type 1 Gaucher disease

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed through Week 41 visit in the TKT025 study.
* Patients must have voluntarily signed an IRB/EC approved informed consent form after all relevant aspects of the study have been explained and discussed with the patient.
* Patient must be sufficiently cooperative to participate in this clinical study as judged by the Investigator.
* Female and male patients of child bearing potential must agree to use a medically acceptable method of contraception at all times during the study. Female patients must have a negative serum pregnancy test on enrollment.

Exclusion Criteria:

* Patient has received treatment with non-Gaucher disease related investigational drug or device within the past 30 days prior to study entry; such use during the study is not permitted.
* Patient has a clinically relevant medical condition (e.g., HIV, hepatitis B or C) that would make implementation of the protocol difficult and/or confound an assessment of the effects of the experimental therapy and its adverse events.
* Patient, patient's parent(s), or patient's legal guardian is unable to understand the nature, scope and possible consequences of the study.
* Patient is unable to comply with the protocol, e.g. uncooperative attitude, medical condition, inability to return for safety evaluations, or is otherwise unlikely to complete the study, as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-09-13 (Actual); Primary Completion 2008-01-31 (Actual); Study Completion 2008-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- Shaare Zedek Medical Center, Jerusalem, Israel
- Maria Sklodowska Curie Children's Hospital, Bucharest, Romania
- Mother and Child Health Care Institute of Serbia, Belgrade, Serbia

REFERENCES:
- [Derived] Zimran A, Altarescu G, Philips M, Attias D, Jmoudiak M, Deeb M, Wang N, Bhirangi K, Cohn GM, Elstein D. Phase 1/2 and extension study of velaglucerase alfa replacement therapy in adults with type 1 Gaucher disease: 48-month experience. Blood. 2010 Jun 10;115(23):4651-6. doi: 10.1182/blood-2010-02-268649. Epub 2010 Mar 18. PMID 20299511

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on 3 February 2005.
Pre-assignment Details: Recruitment of patients was limited to those patient who completed first in man, Phase I/II study TKT025, elected to continue to receive treatment with velaglucerase alfa and met the study inclusion criteria.
Period: Baseline
Arm/Group | GA-GCB
Started | 10
Completed | 10
Not Completed | 0
Period: Month 14
Arm/Group | GA-GCB
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Month 50
Arm/Group | GA-GCB
Started | 9
Completed | 8
Not Completed | 1
Not completed — Physician Decision | 1
Period: Month 84
Arm/Group | GA-GCB
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GA-GCB
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (16.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Serbia | 1
  Israel | 8
  Romania | 1

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Long Term Safety
Description: Overall Summary of Treatment-emergent Adverse Events-Safety Population
Time Frame: Up to 84 months
Population: ITT patient population
Measure: Number; unit: Participants
Groups:
- Number (#) Experienced no Adverse Event (AE): 15-60 U/kg every other week via intravenous infusion
- # Experienced at Least 1 AE; # Experienced at Least 1 Drug-related AE; # Experienced at Least 1 Infusion-related AE; # Experienced at Least 1 Severe AE; # Experienced at Least 1 Drug-related Severe AE; # Experienced at Least 1 Life-threatening AE; # Experienced at Least 1 Serious AE; # Experienced at Least 1 Drug-related Serious AE; # Discontinued Due to an AE: 15-60 U/kg, every other week Intravenously
Arm/Group | Number (#) Experienced no Adverse Event (AE) | # Experienced at Least 1 AE | # Experienced at Least 1 Drug-related AE | # Experienced at Least 1 Infusion-related AE | # Experienced at Least 1 Severe AE | # Experienced at Least 1 Drug-related Severe AE | # Experienced at Least 1 Life-threatening AE | # Experienced at Least 1 Serious AE | # Experienced at Least 1 Drug-related Serious AE | # Discontinued Due to an AE | # Deaths
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
Participants | 0 | 10 | 1 | 1 | 2 | 0 | 0 | 4 | 0 | 0 | 0

2. Secondary Outcome: Percent Change From Baseline in Hemoglobin Concentration
Time Frame: Baseline, then every 12 months
Population: Intent to treat (ITT) patient population
Measure: Mean (Standard Error); unit: Percent Change from Baseline
Groups:
- GA-GCB: 12 Months; GA-GCB: 24 Months; GA-GCB: 36 Months; GA-GCB-48 Months; GA-GCB: 60 Months; GA-GCB: 72 Months; GA-GCB: 84 Months: 15-60 U/kg, every other week Intravenously
Arm/Group | GA-GCB: 12 Months | GA-GCB: 24 Months | GA-GCB: 36 Months | GA-GCB-48 Months | GA-GCB: 60 Months | GA-GCB: 72 Months | GA-GCB: 84 Months
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10
Percent Change from Baseline | 20.91 (1.962) | 20.74 (2.251) | 19.17 (2.365) | 20.96 (3.248) | 16.58 (2.437) | 17.48 (2.317) | 17.97 (2.460)

3. Secondary Outcome: Percent Change From Baseline in Platelet Counts
Time Frame: Baseline, then every 12 months
Population: ITT patient population
Measure: Mean (Standard Error); unit: Percent Change from Baseline
Arm/Group | GA-GCB: 12 Months | GA-GCB: 24 Months | GA-GCB: 36 Months | GA-GCB-48 Months | GA-GCB: 60 Months | GA-GCB: 72 Months | GA-GCB: 84 Months
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10
Percent Change from Baseline | 78.21 (15.127) | 99.60 (15.324) | 111.57 (13.723) | 132.61 (18.461) | 139.73 (27.890) | 126.20 (20.445) | 114.93 (21.783)

4. Secondary Outcome: Percent Change From Baseline in Liver Volume
Time Frame: Baseline, Month 24, then every 9 or 12 months
Population: ITT
Measure: Mean (Standard Error); unit: Percent Change from Baseline
Groups:
- GA-GCB: Month 24; GA-GCB: Month 33; GA-GCB: Month 45; GA-GCB: Month 57; GA-GCB: Month 69; GA-GCB: Month 81: 15-60 U/kg, every other week Intravenously
Arm/Group | GA-GCB: Month 24 | GA-GCB: Month 33 | GA-GCB: Month 45 | GA-GCB: Month 57 | GA-GCB: Month 69 | GA-GCB: Month 81
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Percent Change from Baseline | -28.00 (4.835) | -30.95 (3.627) | -39.35 (4.739) | -38.99 (4.567) | -39.78 (4.821) | -42.07 (4.705)

5. Secondary Outcome: Percent Change From Baseline in Spleen Size
Time Frame: Baseline, Month 24, then every 9 or 12 months
Population: ITT (One patient was excluded due to an intravascular metallic device that prevented accurate spleen evaluation.)
Measure: Mean (Standard Error); unit: Percent Change from Baseline
Arm/Group | GA-GCB: Month 24 | GA-GCB: Month 33 | GA-GCB: Month 45 | GA-GCB: Month 57 | GA-GCB: Month 69 | GA-GCB: Month 81
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
Percent Change from Baseline | -66.86 (6.286) | -68.09 (6.204) | -73.56 (6.717) | -73.97 (6.663) | -75.96 (6.819) | -77.82 (7.002)

ADVERSE EVENTS:
Time Frame: On or after the first infusion in study TK025EXT, up to 7 years.
Arm/Group | GA-GCB
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GA-GCB (N=10)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Scar (Skin and subcutaneous tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (2)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1)
Pyrexia (Gastrointestinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GA-GCB (N=10)
Influenza (Infections and infestations) | 6 (11)
Nasopharyngitis (Infections and infestations) | 5 (5)
Urinary tract infection (Infections and infestations) | 4 (6)
Eye infection (Infections and infestations) | 3 (4)
Nail infection (Infections and infestations) | 2 (2)
Rhinitis (Infections and infestations) | 2 (2)
Acarodermatitis (Infections and infestations) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1)
Fungal rash (Infections and infestations) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Periodontal infection (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (2)
Vaginal infection (Infections and infestations) | 1 (3)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Tinea versicolour (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
vaginal candidiasis (Infections and infestations) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1)
Viral infection (Infections and infestations) | 2 (2)
Condyloma acuminatum (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Asthenopia (Eye disorders) | 1 (1)
Blepharitis (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Eye discharge (Eye disorders) | 1 (1)
Eye inflammation (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1)
Vitreous detachment (Eye disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Hypoacusis (Ear and labyrinth disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (3)
Hypertension (Vascular disorders) | 2 (2)
Haematoma (Vascular disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 7 (19)
Abdominal pain (Gastrointestinal disorders) | 4 (5)
Gingival bleeding (Gastrointestinal disorders) | 4 (6)
Nausea (Gastrointestinal disorders) | 4 (11)
Abdominal discomfort (Gastrointestinal disorders) | 3 (4)
Abdominal pain lower (Gastrointestinal disorders) | 3 (6)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (2)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Scar (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (6)
Groin pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (3)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint crepitation (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spine flattening (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Inflammation (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
Sensation of pressure (General disorders) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1)
Heart rate increased (Investigations) | 1 (1)
Lipids increased (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (4)
Rib fracture (Injury, poisoning and procedural complications) | 2 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 1 (1)
Inguinal hernia repair (Surgical and medical procedures) | 1 (2)
Headache (Nervous system disorders) | 6 (10)
Dizziness (Nervous system disorders) | 3 (12)
Hypoaesthesia (Nervous system disorders) | 2 (4)
Paraesthesia (Nervous system disorders) | 2 (2)
Aphasia (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Circadian rhythm sleep disorder (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Muscle Spasticity (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1)
Cervix disorder (Reproductive system and breast disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1)
Premenstrual syndrome (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Pyrexia (General disorders) | 6 (7)
Fatigue (General disorders) | 5 (5)
Asthenia (General disorders) | 3 (3)
Malaise (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 2 (4)
Adverse drug reaction (General disorders) | 1 (1)
Feeling hot (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Imputation was applied to missing data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Shire's agreements with investigators vary. All agreements provide Shire the right to embargo communications regarding trial results prior to public release for a period ≤180 days from the time submitted to Shire for review. Shire does not prohibit publication, but can require the removal of confidential information (excluding trial results) and can request postponement of a single-center publication until after disclosure of the trial's multi-center publication.